CLINICAL TRIAL: NCT00204451
Title: Human Ovarian Follicular Dynamics and Emergency Contraception
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Roger Pierson, Ph.D., FEAS, FCAHS, MS, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Bio 05-67; CIHR MOP 11489
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Contraception
Keywords: emergency contraception; follicle; ovulation; blood pressure; Fertility Control; Inhibition of fertilization

INTERVENTIONS:
Drug: 0.75 levonorgestrel
Drug: 50 mg ethinyl estradiol/0.5 mg levonorgestrel

SUMMARY:
The researchers hypothesize that emergency contraception (EC) will initiate the changes associated with atresia or ovulatory failure at all stages of follicular development and that the image attributes associated with atresia will be similar regardless of the diameter of the dominant follicle when ovarian suppression is initiated. Second, changes associated with atresia may be observed, but ovulation of the dominant follicle is unimpeded.

DETAILED DESCRIPTION:
This study is a single-center, randomized, open-label, double-controlled protocol to study the pattern of ovarian follicular growth and regression in two groups of women. The first group will use Plan B, which is a progesterone only OC containing 0.75 levonorgestrel. The second group of women will use the Yuzpe regimen, which uses 50 mg ethinyl estradiol/0.5 mg levonorgestrel pills at different stages of the menstrual follicular cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Female volunteers of childbearing potential;
2. Are first time users of oral contraception (OC) or have discontinued OC at least 1 month prior to study entry;
3. Age between 18 and 40 years old;
4. Normal body mass index (18-38);
5. Has signed informed consent form; and
6. Is in good health as confirmed by medical history, physical examination.

Exclusion Criteria:

1. A positive pregnancy test will automatically exclude the volunteer from participation in this study.
2. Any contraindication for oral contraception use;
3. Irregular menstrual cycles;
4. Ultrasonographic evidence of ovarian dysfunction, such as polycystic ovary syndrome (PCOS);
5. Pregnancy (suspected or diagnosed) or lactation;
6. History or suspicion of drug or alcohol abuse;
7. Participation in an investigational drug trial within the 30 days prior to selection;
8. Exhibits a disorder that is a contraindication to steroid hormonal therapy, including, for example, the following conditions:

   * history of, or actual, thrombophlebitis or thromboembolic disorders.
   * history of, or actual, cerebrovascular disorders.
   * history of, or actual, myocardial infarction or coronary artery disease.
   * acute liver disease.
   * history of, or actual, benign or malignant liver tumors.
   * history of, or suspected, carcinoma of the breast.
   * known, or suspected, estrogen-dependent neoplasia.
   * undiagnosed abnormal vaginal bleeding.
   * any ocular lesion arising from ophthalmic vascular disease, such as partial or complete loss of vision or defect in visual field.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Start 2005-07; Study Completion 2006-06

PRIMARY OUTCOMES:
follicle development
ovulation status
peripheral blood pressure

SECONDARY OUTCOMES:
endometrial development

CONTACTS AND LOCATIONS:
Overall Officials: Roger A Pierson, MS PhD, Principal Investigator — University of Saskatchewan; Salma T Hanna, MD PhD, Study Director — University of Saskatchewan; Olufemi A Olatunbosun, MD, Study Chair — University of Saskatchewan
Locations (1):
- Ob-Gyn Royal University Hospital, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Background] Pierson RA, Archer DF, Moreau M, Shangold GA, Fisher AC, Creasy GW. Ortho Evra/Evra versus oral contraceptives: follicular development and ovulation in normal cycles and after an intentional dosing error. Fertil Steril. 2003 Jul;80(1):34-42. doi: 10.1016/s0015-0282(03)00556-9. PMID 12849799
- [Background] Baerwald AR, Adams GP, Pierson RA. A new model for ovarian follicular development during the human menstrual cycle. Fertil Steril. 2003 Jul;80(1):116-22. doi: 10.1016/s0015-0282(03)00544-2. PMID 12849812